CLINICAL TRIAL: NCT00778700
Title: A Double-Blind, Randomized, Vehicle-Controlled Dose Ranging Study of the Effect of INCB018424 Phosphate Cream When Applied to Patients With Plaque Psoriasis
Brief Title: A Dose Ranging Study of the Effect of Ruxolitinib Phosphate Cream When Applied to Participants With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 18424-203
Record Dates: First submitted 2008-10-21; First posted 2008-10-23 (Estimated); Results first posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (4):
- Vehicle Cream (Placebo Comparator): Vehicle cream, applied topically, once daily from Day 1 to Week 12.
  Interventions: Other: Placebo Cream
- Ruxolitinib Phosphate 0.5% Cream (Experimental): Ruxolitinib phosphate 0.5% cream, applied topically, once daily from Day 1 to Week 12.
  Interventions: Drug: Ruxolitinib Phosphate
- Ruxolitinib Phosphate 1.0% Cream (Experimental): Ruxolitinib phosphate 1.0% cream, applied topically, once daily from Day 1 to Week 12.
  Interventions: Drug: Ruxolitinib Phosphate
- Ruxolitinib Phosphate 1.5% Cream (Experimental): Ruxolitinib phosphate 1.5% cream, applied topically, once daily from Day 1 to Week 12.
  Interventions: Drug: Ruxolitinib Phosphate

INTERVENTIONS:
Other: Placebo Cream — Cream with no active drug
  Arms: Vehicle Cream
Drug: Ruxolitinib Phosphate — Ruxolitinib phosphate cream
  Other Names: INCB018424
  Arms: Ruxolitinib Phosphate 0.5% Cream; Ruxolitinib Phosphate 1.0% Cream; Ruxolitinib Phosphate 1.5% Cream

SUMMARY:
The study was double-blind, randomized, vehicle-controlled study with application of Ruxolitinib phosphate cream or vehicle cream in participants with stable plaque psoriasis applied once daily for 12 weeks without occlusive dressings. There were 4 treatment groups anticipated to have 50 participants in each.

ELIGIBILITY:
Inclusion Criteria:

* Plaque psoriasis involving up to 2 to 20% Body Surface Area

Exclusion Criteria:

* Lesions solely involving intertriginous areas, the scalp or the face
* Systemic therapy for their psoriasis
* Pustular psoriasis or erythroderma
* Currently on other topical agents or Ultraviolet B (UVB) therapy within 2 weeks of the first dose of study medication
* Started or discontinued therapy within 2 months of Screening with agents that can exacerbate psoriasis
* Receiving systemic triazole antifungals except fluconazole

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2008-10-28 (Actual); Primary Completion 2009-06-26 (Actual); Study Completion 2009-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Luchi, M.D., Study Director — Incyte Corporation
Locations (28):
- United States (28):
  - Hot Springs, Arkansas
  - Los Angeles, California
  - San Diego, California
  - Santa Monica, California
  - Vallejo, California
  - New Haven, Connecticut
  - Miami, Florida
  - Ormond Beach, Florida
  - Naperville, Illinois
  - Wheaton, Illinois
  - Evansville, Indiana
  - South Bend, Indiana
  - Boston, Massachusetts
  - Clinton Township, Michigan
  - Fridley, Minnesota
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - Rochester, New York
  - Norman, Oklahoma
  - Simpsonville, South Carolina
  - Austin, Texas
  - College Station, Texas
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Walla Walla, Washington
  - Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 199 participants were enrolled at 27 sites in the United States from 28 October 2008 to 26 June 2009.
Pre-assignment Details: 220 participants with stable plaque psoriasis were enrolled in the study, 199 of whom received randomized study drug and were analyzed in this study. 21 subjects did not receive study drug and were therefore excluded from the ITT and Safety analysis sets. The participants were randomized in 1:1:1:1 ratio to receive vehicle cream or Ruxolitinib phosphate 0.5% cream or Ruxolitinib phosphate 1.0% cream or Ruxolitinib phosphate 1.5% cream.
Period: Overall Study
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Started | 50 | 51 | 49 | 49
Completed | 32 | 44 | 43 | 36
Not Completed | 18 | 7 | 6 | 13
Not completed — Adverse Event | 6 | 1 | 3 | 5
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Subject Withdrew Consent | 6 | 4 | 1 | 4
Not completed — Lost to Follow-up | 3 | 1 | 0 | 1
Not completed — Reason not Specified | 2 | 0 | 1 | 3
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were enrolled and used at least one application of study drug.
Groups:
- Vehicle: Vehicle cream, applied topically, once daily from Day 1 to Week 12.
- Total: Total of all reporting groups
Arm/Group | Vehicle | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream | Total
Number analyzed (Participants) | 50 | 51 | 49 | 49 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (10.94) | 45.4 (10.91) | 44.9 (13.03) | 43.6 (12.80) | 44.0 (11.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 24 | 23 | 84
  Male | 33 | 31 | 25 | 26 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 8 | 3 | 26
  Not Hispanic or Latino | 41 | 45 | 41 | 46 | 173
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian Native | 45 | 46 | 46 | 48 | 185
  Black or African American | 2 | 2 | 1 | 1 | 6
  Asian | 1 | 0 | 1 | 0 | 2
  Other | 2 | 3 | 1 | 0 | 6
Total Lesion Score [Mean (Full Range); unit: score on a scale] — Total Lesion Score is calculated as the sum of component scores for erythema (E), scaling (S), and thickness (T) of the study-treated lesions taken together. Each component score can vary in value from 1 to 12. A negative change from Baseline indicates improvement.
  All participants who were randomized to treatment and had both a baseline visit and received at least one application of study drug were included in the Intent-to-Treat (ITT) population.
  score on a scale | 7.2 [5 to 11] | 7.1 [5 to 10] | 6.7 [5 to 11] | 7.1 [5 to 12] | 7.0 [5 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Total Lesion Score for All Treatable Psoriatic Lesions to Day 84
Description: Total Lesion Score is calculated as the sum of component scores for erythema (E), scaling (S), and thickness (T) of the study-treated lesions taken together. Each component consists of ratings of 0=none, 1=mild, 2=moderate, 3=marked, and 4=severe such that total lesion score can vary in value from 0 to 12. A negative change from Baseline indicates improvement.
Time Frame: From Baseline (Day 1) to Day 84
Population: All participants who were randomized to treatment and had both a baseline visit and received at least one application of study drug were included in the ITT population. Overall number of participants analyzed are the participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Number analyzed (Participants) | 47 | 49 | 49 | 48
score on a scale | -1.07 (0.290) | -2.25 (0.284) | -2.47 (0.285) | -2.27 (0.287)
Statistical Analysis 1: Comparison: Vehicle Cream vs Ruxolitinib Phosphate 0.5% Cream; Test type: Superiority; p = 0.0041, ANCOVA; The ANCOVA model included treatment as the main factor and Baseline score as the covariate; Least Squares (LS) Mean Difference = -1.18, 90% CI 2-sided [-1.85 to -0.51], Standard Error of Mean 0.406
Statistical Analysis 2: Comparison: Vehicle Cream vs Ruxolitinib Phosphate 1.0% Cream; Test type: Superiority; p = 0.0007, ANCOVA; The ANCOVA model included treatment as the main factor and Baseline score as the covariate; LS Mean Difference = -1.40, 90% CI 2-sided [-2.08 to -0.73], Standard Error of Mean 0.408
Statistical Analysis 3: Comparison: Vehicle Cream vs Ruxolitinib Phosphate 1.5% Cream; Test type: Superiority; p = 0.0035, ANCOVA; The ANCOVA model included treatment as the main factor and Baseline score as the covariate; LS Mean Difference = -1.21, 90% CI 2-sided [-1.88 to -0.53], Standard Error of Mean 0.407

2. Secondary Outcome: Absolute Change From Baseline in the Individual Lesion Scores for Lesion Thickness
Description: Lesion thickness was scored using a 5-point scale ranging from 0 to 4 where 0 is none or absent and 4 is severe lesion. A negative change from Baseline indicates improvement.
Time Frame: From Baseline (Day 1) to Day 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Number analyzed (Participants) | 47 | 49 | 48 | 48
score on a scale | -0.45 (0.775) | -0.71 (0.677) | 0.84 (0.898) | -0.90 (0.778)

3. Secondary Outcome: Absolute Change From Baseline in the Individual Lesion Scores for Lesion Erythema
Description: Lesion erythema was scored using a 5-point scale ranging from 0 to 4 where 0 is none or absent and 4 is severe lesion. A negative change from Baseline indicates improvement.
Time Frame: From Baseline (Day 1) to Day 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Number analyzed (Participants) | 33 | 44 | 45 | 39
score on a scale | -0.45 (0.711) | -0.59 (0.757) | -0.72 (0.889) | -0.64 (0.872)

4. Secondary Outcome: Absolute Change From Baseline in the Individual Lesion Scores for Lesion Scaling
Description: Lesion scaling was scored using a 5-point scale ranging from 0 to 4 where 0 is none or absent and 4 is severe lesion. A negative change from Baseline indicates improvement.
Time Frame: From Baseline (Day 1) to Day 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Number analyzed (Participants) | 33 | 44 | 45 | 39
score on a scale | -0.46 (0.972) | -0.91 (0.741) | -0.87 (0.991) | -0.85 (0.961)

5. Secondary Outcome: Percent Change From Baseline in the Individual Lesion Scores of Lesion Thickness
Description: Lesion thickness was scored using a 5-point scale ranging from 0 to 4 where 0 is none or absent and 4 is severe lesion. A negative percent change from Baseline indicates improvement in lesion.
Time Frame: From Baseline (Day 1) to Day 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Number analyzed (Participants) | 47 | 49 | 49 | 48
percent change | -17.37 (31.075) | -30.95 (27.851) | -36.56 (38.447) | -36.80 (33.016)

6. Secondary Outcome: Percent Change From Baseline in the Individual Lesion Scores of Lesion Erythema
Description: Lesion erythema was scored using a 5-point scale ranging from 0 to 4 where 0 is none or absent and 4 is severe lesion. A negative percent change from Baseline indicates improvement in lesion.
Time Frame: From Baseline (Day 1) to Day 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Number analyzed (Participants) | 33 | 44 | 45 | 39
percent change | -15.40 (22.146) | -22.53 (27.702) | -30.74 (39.404) | -23.93 (35.828)

7. Secondary Outcome: Percent Change From Baseline in the Individual Lesion Scores of Lesion Scaling
Description: Lesion scaling was scored using a 5-point scale ranging from 0 to 4 where 0 is none or absent and 4 is severe lesion. A negative percent change from Baseline indicates improvement in lesion.
Time Frame: From Baseline (Day 1) to Day 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Number analyzed (Participants) | 33 | 44 | 45 | 39
percent change | -17.68 (38.175) | -37.13 (28.050) | -35.38 (44.140) | -36.11 (41.286)

8. Secondary Outcome: Percentage of Participants Achieving None (Score=0) and Mild (Score=1) in Lesion Thickness at Day 84
Description: Lesion thickness was scored using a 5-point scale ranging from 0 to 4 where 0 is none or absent and 4 is severe lesion. Participants with individual lesion scores 0 (none) and 1 (mild) are reported in this outcome measure.
Time Frame: Day 84
Population: All participants who were randomized to treatment and had both a baseline visit and received at least one application of study drug were included in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Number analyzed (Participants) | 50 | 51 | 49 | 49
percentage of participants | 25.5 | 55.1 | 55.1 | 50.0

9. Secondary Outcome: Percentage of Participants Achieving None (Score=0) and Mild (Score=1) in Lesion Erythema at Day 84
Description: The individual lesion scores were calculated individually for thickness, erythema, and scaling. Lesion erythema was scored using a 5-point scale ranging from 0 to 4 where 0 is none or absent and 4 is severe lesion. Participants with individual lesion scores 0 (none) and 1 (mild) are reported in this outcome measure. The LOCF method was used for analysis.
Time Frame: Day 84
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Number analyzed (Participants) | 50 | 51 | 49 | 49
percentage of participants | 19.1 | 34.7 | 46.9 | 33.3

10. Secondary Outcome: Percentage of Participants Achieving None (Score=0) and Mild (Score=1) in Lesion Scaling at Day 84
Description: The individual lesion scores were calculated individually for thickness, erythema, and scaling. Lesion scaling was scored using a 5-point scale ranging from 0 to 4 where 0 is none or absent and 4 is severe lesion. Participants with individual lesion scores 0 (none) and 1 (mild) are reported in this outcome measure. The LOCF method was used for analysis.
Time Frame: Day 84
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Number analyzed (Participants) | 50 | 51 | 49 | 49
percentage of participants | 42.6 | 61.2 | 63.3 | 50.0

11. Secondary Outcome: Absolute Change From Baseline in the Percent Treatable Body Surface Area (BSA)
Description: The lesion areas were estimated based on the Rule of Nines method for the entire skin surface; psoriatic disease activity and the percent BSA were calculated for the treatable areas (i.e., areas that excluded the scalp, face, and intertriginous areas). The BSA is calculated as follows: BSA (m^²)=([Height(cm) x Weight(kg)]/3600 )^½. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Day 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent treatable BSA
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Number analyzed (Participants) | 47 | 49 | 49 | 48
Percent treatable BSA | -0.36 (2.260) | -1.63 (3.746) | -2.41 (4.276) | -1.94 (3.545)

12. Secondary Outcome: Absolute Change From Baseline in the Physician's Global Assessment (PGA) Score
Description: The overall disease activity in the participants, a measure of the overall quality (erythema, scaling, and thickness) and extent (BSA) of plaques, was measured using the PGA. The PGA was an overall assessment of each participant's plaque psoriasis. The assessment was recorded using a 6-point scale ranging from 0 to 5 where 0 is 'Clear' (no evidence of disease) and 5 is 'very Severe' lesion. A negative change from Baseline indicates improvement. The ANCOVA method was used for analyses.
Time Frame: Baseline (Day 1) to Day 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Number analyzed (Participants) | 47 | 49 | 48 | 48
score on a scale | -0.34 (0.760) | -0.73 (0.836) | -0.92 (1.077) | -0.79 (0.922)

13. Secondary Outcome: Percent Change From Baseline in the PGA Score
Description: The overall disease activity in the participants, a measure of the overall quality (erythema, scaling, and thickness) and extent (BSA) of plaques, was measured using the PGA. The PGA was an overall assessment of each participant's plaque psoriasis. The assessment was recorded using a 6-point scale ranging from 0 to 5 where 0 indicates 'Clear' (no evidence of disease) and 5 indicates 'very Severe' lesion. A negative percent change indicates improvement. The ANCOVA method was used for analyses.
Time Frame: Baseline (Day 1) to Day 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Number analyzed (Participants) | 47 | 49 | 49 | 47
percent change from baseline | -9.09 (23.624) | -22.10 (24.626) | -29.69 (34.344) | -23.33 (26.485)

14. Secondary Outcome: Percentage of Participants Achieving Clear (Score=0) and Almost Clear (Score=1) on the PGA
Description: The overall disease activity in the participants, a measure of the overall quality (erythema, scaling, and thickness) and extent (BSA) of plaques, was measured using the PGA. The PGA was an overall assessment of each participant's plaque psoriasis. The assessment was recorded using a 6-point scale ranging from 0 to 5 where 0 indicates 'Clear' (no evidence of disease) and 5 indicates 'very Severe' lesion. Participants with individual lesion scores 0 (clear) and 1 (almost clear) are reported in this outcome measure.
Time Frame: Day 84
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Number analyzed (Participants) | 50 | 51 | 49 | 49
percentage of participants | 4.3 | 12.2 | 32.7 | 12.5

15. Secondary Outcome: Absolute Change From Baseline in the Psoriasis Area and Severity Index (PASI) Score
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring [lower extremities, trunk (including stomach, chest, back), upper extremities, head]; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by scale 0 (none) to 4 (severe). Final PASI is the sum of severity score for each area multiplied coverage for each section multiplied by area score weight of section (lower extremities: 0.4, trunk: 0.3, upper extremities: 0.2, head: 0.1). A negative change from baseline indicates improvement. The ANCOVA method was used for analyses.
Time Frame: Baseline (Day 1) to Day 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Number analyzed (Participants) | 47 | 49 | 49 | 48
score on a scale | -1.49 (2.999) | -3.47 (3.951) | -3.48 (4.204) | -2.93 (3.599)

16. Secondary Outcome: Percent Change From Baseline in the PASI Score
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring [lower extremities, trunk (including stomach, chest, back), upper extremities, head]; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by scale 0 (none) to 4 (severe). Final PASI is the sum of severity score for each area multiplied by coverage for each section multiplied by area score weight of section (lower extremities: 0.4, trunk: 0.3, upper extremities: 0.2, head: 0.1). A percent negative change from baseline indicates improvement in disease. The ANCOVA method was used for analyses.
Time Frame: Baseline (Day 1) to Day 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Number analyzed (Participants) | 47 | 49 | 49 | 48
percent change | -18.45 (29.907) | -34.19 (40.532) | -39.97 (38.215) | -32.81 (38.995)

17. Secondary Outcome: Percentage of Participants With Treatable Percent BSA ≥10% Achieving PASI 50%, PASI 75%, And PASI 90% Improvements From Baseline to Each Time Point
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring [lower extremities, trunk (including stomach, chest, back), upper extremities, head]; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by scale 0 (none) to 4 (severe). Final PASI is the sum of severity score for each area* multiplied by coverage for each section* multiplied by area score weight of section (lower extremities: 0.4, trunk: 0.3, upper extremities: 0.2, head: 0.1). A negative percent change from Baseline indicates improvement. Data for Day 84 was imputed using the LOCF method.
Time Frame: Baseline (Day 1) and Days 15, 28, 56, 84, and 112
Population: All participants who were randomized to treatment and had both a baseline visit and received at least one application of study drug were included in the ITT population. Overall number analyzed are the participants with percent treatable BSA of at least 10%.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Number analyzed (Participants) | 18 | 11 | 20 | 17
percentage of participants
  Achieved 50% Reduction on Day 15 | 0.0 | 0.0 | 20.0 | 18.8
  Achieved 50% Reduction on Day 28 | 0.0 | 11.1 | 33.3 | 25.0
  Achieved 50% Reduction on Day 56 | 16.7 | 50.0 | 21.1 | 38.5
  Achieved 50% Reduction on Day 84 | 18.8 | 60.0 | 45.0 | 37.5
  Achieved 50% Reduction on Day 112 | 17.6 | 66.7 | 31.6 | 17.6
  Achieved 75% Reduction on Day 15 | 0.0 | 0.0 | 5.0 | 0.0
  Achieved 75% Reduction on Day 28 | 0.0 | 0.0 | 5.6 | 0.0
  Achieved 75% Reduction on Day 56 | 0.0 | 25.0 | 10.5 | 7.7
  Achieved 75% Reduction on Day 84 | 0.0 | 30.0 | 15.0 | 12.5
  Achieved 75% Reduction on Day 112 | 0.0 | 33.3 | 15.8 | 11.8
  Achieved 90% Reduction on Day 15 | 0.0 | 0.0 | 0.0 | 0.0
  Achieved 90% Reduction on Day 28 | 0.0 | 0.0 | 0.0 | 0.0
  Achieved 90% Reduction on Day 56 | 0.0 | 0.0 | 5.3 | 7.7
  Achieved 90% Reduction on Day 84 | 0.0 | 0.0 | 15.0 | 6.3
  Achieved 90% Reduction on Day 112 | 0.0 | 0.0 | 15.8 | 5.9

18. Secondary Outcome: Trough Plasma Concentrations [Minimum Concentration at Steady-state (Css,Min)] of Ruxolitinib Phosphate Prior to Study Drug Application at Steady State
Time Frame: Pre-application on Days 1, 15, 28, 56, and 84
Population: All participants who used at least one application of study medication, and provided at least one plasma sample were considered potentially evaluable for the pharmacokinetic (PK)/ pharmacodynamic (PD) population.
Measure: Mean (Standard Deviation); unit: nanomolar (nM)
Arm/Group | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream
Number analyzed (Participants) | 51 | 49 | 49
nanomolar (nM) | 9.19 (11.77) | 16.99 (19.05) | 19.97 (25.13)

ADVERSE EVENTS:
Time Frame: From first dose up to 28 days after last dose of study drug (Up to 16 weeks)
Description: Safety population included all participants who were enrolled and used at least one application of study drug.
Groups:
- Vehicle Cream: Vehicle cream Vehicle cream, applied topically, once daily from Day 1 to Week 12.
- Total: Total
Arm/Group | Vehicle Cream | Ruxolitinib Phosphate 0.5% Cream | Ruxolitinib Phosphate 1.0% Cream | Ruxolitinib Phosphate 1.5% Cream | Total
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51 | 0/49 | 0/49 | 0/199
Serious Adverse Events (participants affected / at risk) | 1/50 | 2/51 | 0/49 | 3/49 | 6/199
Other Adverse Events (participants affected / at risk) | 11/50 | 11/51 | 16/49 | 18/49 | 56/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Cream (N=50) | Ruxolitinib Phosphate 0.5% Cream (N=51) | Ruxolitinib Phosphate 1.0% Cream (N=49) | Ruxolitinib Phosphate 1.5% Cream (N=49) | Total (N=199)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Cream (N=50) | Ruxolitinib Phosphate 0.5% Cream (N=51) | Ruxolitinib Phosphate 1.0% Cream (N=49) | Ruxolitinib Phosphate 1.5% Cream (N=49) | Total (N=199)
Application site irritation (General disorders) | 3 (3) | 1 (2) | 2 (2) | 5 (6) | 11 (13)
Application site pruritus (General disorders) | 4 (5) | 2 (3) | 2 (2) | 2 (2) | 10 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 5 (5)
Electrocardiogram QT interval abnormal (Investigations) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 5 (5)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (16) | 1 (2) | 4 (18)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 6 (6)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (3) | 3 (3) | 5 (5) | 11 (12)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 6 (8) | 1 (1) | 3 (3) | 13 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.